CLINICAL TRIAL: NCT04920240
Title: Application of Multi-center Unified High-frequency Contact Surface Standardized Cleaning and Disinfection Mode in Hospital Infection Prevention and Control in ICU
Brief Title: Application of Standardized Cleaning and Disinfection Mode of HFT Surface in Hospital Infection Prevention and Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Jiaxing University (Other); Changxing People's Hospital (Other); Yuhang Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2020-203
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-05

CONDITIONS: Hospital Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Multi-center unification, before-after study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine group (Placebo Comparator): In accordance with the "intensive care unit hospital infection prevention and control norms" requirements
  Interventions: Behavioral: Routine procedure
- Experimental group (Experimental): Implement a multi-center unified ICU high-frequency contact surface standardized cleaning and disinfection mode
  Interventions: Behavioral: cleaning and disinfection mode for surfaces with high frequency contact

INTERVENTIONS:
Behavioral: cleaning and disinfection mode for surfaces with high frequency contact — According to the results of the survey on the status of high frequency contact surface, the corresponding frequency and method of cleaning and disinfection are determined. Set up a multidisciplinary quality control team.
  Arms: Experimental group
Behavioral: Routine procedure — clean the high frequency contact surface like other surfaces
  Arms: routine group

SUMMARY:
The scientific, feasible and effective mode of standardized cleaning and disinfection of ICU high-frequency contact surfaces is discussed and verified.

DETAILED DESCRIPTION:
This study is a multi-center unified interventional study, using the front and rear control method, it is proposed to improve the ICU traditional cleaning and disinfection method on the basis of the ICU high-frequency contact surface status survey, explore the best frequency and disinfection method of ICU high-frequency contact surface cleaning and disinfection, establish a multi-center unified ICU high-frequency contact surface standardized cleaning and disinfection mode, in order to achieve the ideal cleaning and disinfection effect, effective prevention and control of ICU hospital infection occurrence and transmission.

ELIGIBILITY:
Inclusion Criteria:

* High-frequency contact with the surface of an object by ICU patients and their surroundings; informed consent.

Exclusion Criteria:

* Admission < 24 hours; < 18 years old; hospital infection prior to admission to the ICU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital infections | 1 year
  the difference of Incidence of hospital infections

CONTACTS AND LOCATIONS:
Overall Officials: Jiangshuyuan Liang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No